CLINICAL TRIAL: NCT00339001
Title: The Possible Influence of Erythropoietin and Early Iron Supplements on the Prevalence and Severity of Retinopathy of Prematurity and Other Short Term Outcome of Prematurity
Brief Title: Erythropoietin and Early Iron Supplement and Retinopathy of Prematurity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-06-4128-JK-CTIL
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Last update posted 2006-06-20 (Estimated); Status verified 2006-06

CONDITIONS: Retinopathy of Prematurity
Keywords: Erythropoietin; Iron; Retinopathy of prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Erythropoietin

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

INTERVENTIONS:
Drug: erythropoietin and early iron supplements

SUMMARY:
To evaluate the possibility that erythropoietin with early iron supplementation may induce retinopathy of prematurity or worsen this disease. In addition risk factors for the development of ROP will be checked.

ELIGIBILITY:
Inclusion Criteria:

* all premature infants with birth weight of 1250 grams or less

Exclusion Criteria:

* none

Ages: 2 Weeks to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400
Dates: Start 2006-04; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Kuint, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Neonatal Department, Sheba Medical Center, Ramat Gan, Israel